CLINICAL TRIAL: NCT00001601
Title: Patient Evaluation and Treatment of Oral Soft Tissue Diseases According to Generally Available, Standard Procedures and Therapeutic Modalities
Brief Title: Evaluation and Treatment of Oral Soft Tissue Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970169; 97-D-0169
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-08

CONDITIONS: Aphthous Stomatitis; Burning Mouth Syndrome; Lichen Planus; Mouth Disease; Temporomandibular Joint Disorder
Keywords: Oral Medicine; Clinical Experience; Therapy; Educational Training; Pathogenesis; Oral Lesions; Aphthous Ulcers; Lichen Planus; Burning Mouth; Temporomandibular Dysfunction (TMD); Oral Disease; Oral Manifestations
MeSH Terms: conditions — Stomatitis, Aphthous; Burning Mouth Syndrome; Lichen Planus; Mouth Diseases; Temporomandibular Joint Disorders; Oral Manifestations | interventions — Biopsy; X-Rays

INTERVENTIONS:
Procedure: Electrocardiogram
Procedure: Biopsies
Procedure: Diagnostic imaging

SUMMARY:
This study offers evaluation and treatment of patients with diseases of the mouth or systemic diseases that involve the mouth. The protocol is not designed to test new treatments; rather, patients will receive current standard of care treatments. The purposes of the study are: 1) to allow NIDCR's Gene Therapy and Therapeutics Branch staff to gain more knowledge about oral soft tissue diseases and possibly identify new avenues of research in this area; and 2) to establish a pool of patients who may be eligible for new studies as they are developed. (Participants in this protocol will not be required to join a new study; the decision will be voluntary.)

Patients of any age with oral diseases or systemic diseases involving the mouth may be eligible for this study. Women of childbearing potential and women who are pregnant or breastfeeding will only have tests and procedures and receive medications that pose no greater than a minimal risk to the fetus.

Participants will have a comprehensive dental and medical examination, including a physical examination of the head and neck. Additional tests and procedures that may be required for diagnosis and to guide treatment include the following:

* Blood and urine tests - for routine laboratory studies, assessment of kidney and liver function, and detection of viruses, fungi, bacteria or parasites
* Electrocardiogram - to record the electrical activity of the heart
* Biopsies - to examine tissue under the microscope. The method and number of biopsies depends on the individual's specific condition and the tissue to be removed. For all biopsies a local anesthetic (lidocaine with or without epinephrine) is injected at the biopsy site. A punch biopsy uses a small sharp cookie-cutter instrument to remove a small (about 1/10- to 1/5-inch) piece of skin. An excisional biopsy uses a small surgical knife or scalpel to remove a piece of tissue, usually requiring some stitches to close the wound.
* Diagnostic imaging - X-rays, photographs, or other tests as needed for diagnosis

Treatments include tablets, injections and topically applied medications. All preparations are approved by the Food and Drug Administration and are commercially available. Patient follow-up may vary from one visit to intermittent visits over a number of years, depending on the patient's condition.

DETAILED DESCRIPTION:
The function of this protocol is to support the training of residents in Oral Medicine in the management of oral soft tissue diseases. Patients enrolled in this protocol will be evaluated and treated according to available standard procedures and therapeutic modalities. Samples of blood and oral tissues will be studied by routine and specialized investigative methods to establish the diagnoses, responses to treatment, and/or disease progression.

ELIGIBILITY:
INCLUSION CRITERIA

Patients of any age, both genders, and all racial/ethnic groups with oral diseases or systemic diseases with oral manifestations that will help the branch fulfill the objectives listed in Section 1.0.

Women of childbearing potential, or who are pregnant or lactating, will only undergo tests and procedures, and/or receive medications for which data exists proving minimal risk to the fetus and/or child. Only diagnosis without radiographs will be performed.

EXCLUSION CRITERIA

A written referral is needed from the patient's physician or dentist.

No patients with significant cognitive impairment.

No pregnancy or lactation, if this status precludes proposed diagnostic procedures or therapies because of unknown, untoward effects on mother and/or child.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 999
Dates: Start 1997-08; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lozada-Nur F, Miranda C. Oral lichen planus: epidemiology, clinical characteristics, and associated diseases. Semin Cutan Med Surg. 1997 Dec;16(4):273-7. doi: 10.1016/s1085-5629(97)80016-8. PMID 9421218
- [Background] Axell T, Pindborg JJ, Smith CJ, van der Waal I. Oral white lesions with special reference to precancerous and tobacco- related lesions: conclusions of an international symposium held in Uppsala, Sweden, May 18-21 1994. International Collaborative Group on Oral White Lesions. J Oral Pathol Med. 1996 Feb;25(2):49-54. doi: 10.1111/j.1600-0714.1996.tb00191.x. PMID 8667255
- [Background] Ship JA. Recurrent aphthous stomatitis. An update. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Feb;81(2):141-7. doi: 10.1016/s1079-2104(96)80403-3. PMID 8665304